CLINICAL TRIAL: NCT06239870
Title: Single-arm, Single-center, Exploratory Phase II Clinical Study of Envafolimab Combined With Chemoradiotherapy in the Treatment of Locally Advanced pMMR/MSS Rectal Cancer
Acronym: ESTIMATE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yunnan Cancer Hospital (Other)
Collaborators: Beijing Bethune Charitable Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLKYLX2023-006; STLKY0036 (Other Grant/Funding Number: Beijing Bethune Public Welfare Foundation)
Record Dates: First submitted 2024-01-03; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Envafolimab Combined With Chemoradiotherapy in the Treatment of Locally Advanced pMMR/MSS Rectal Cancer
Keywords: Local progressive stage; Rectal cancer; Full neoadjuvant therapy; pMMR/MSS; Envafolimab
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant therapy (Experimental): 1. Induction therapy stage: chemotherapy combined with immunotherapy for 2 cycles: Envafolimab: 200mg, subcutaneous injection, Q2W, 2 cycles; mFOLFOX6: Q2W, 2 cycles (concurrent administration of envollizumab on the first day of chemotherapy).
  2. Concurrent chemoradiotherapy: long-term chemoradiotherapy combined with immunotherapy for 3 cycles: radiation therapy: 50Gy/25f, 2Gy every day, 5 days a week for 5 weeks; Capecitabine: 825mg/m2 orally (1650mg/m2/d) twice a day in the morning and evening, 5 days a week, simultaneous with radiation therapy, for a total of 25 days; Envafolimab: 200mg, subcutaneous injection, Q2W, 3 cycles (Envafolimab was administered on day 1, day 15, and day 29 of radiotherapy).
  Iii. Consolidation treatment stage: chemotherapy combined with immunotherapy for 2 cycles: Envafolimab: 200mg, subcutaneous injection, Q2W, 2 cycles; mFOLFOX6: Q2W, 2 cycles. (Concurrent administration of envafolimab on the first day of chemotherapy).
  Interventions: Drug: Envafolimab combined with chemoradiotherapy in the whole course of neoadjuvant therapy

INTERVENTIONS:
Drug: Envafolimab combined with chemoradiotherapy in the whole course of neoadjuvant therapy — Each enrolled patient was given 2 cycles of induction chemotherapy combined with immunization, followed by immunization combined with chemoradiotherapy, and finally 2 cycles of consolidation chemotherapy combined immunization

SUMMARY:
Preoperative radiotherapy combined with 5-fluorouracil/capecitabine is currently the standard treatment for locally advanced rectal cancer. Although this strategy effectively reduces the risk of local recurrence, it fails to effectively improve the overall survival rate of patients . The root cause is that 5-fluorouracil/capecitabine based local radiotherapy is not effective in controlling potential micrometastases. Therefore, many studies try to combine preoperative radiotherapy with more intense chemotherapy and targeted drugs at the same time, as well as induction chemotherapy before preoperative radiotherapy and consolidation chemotherapy after, in order to obtain better efficacy. However, a number of studies have shown that increasing cytotoxic drugs fail to effectively improve pathologic complete response rate (pCR) and long-term survival rate, and significantly increase therapeutic toxicity . Therefore, the idea of trying to increase the efficacy of cytotoxic drugs by accumulating them does not work.Based on the use of PD-1/PD-L1 antibody in colorectal cancer and other solid tumors, and referring to the scheme of PD-1/PD-L1 antibody combined with radiotherapy in other solid tumors, we added envafolimab to local radiotherapy for advanced rectal cancer for exploration, with a view to further improving the pCR rate and long-term survival of patients.

DETAILED DESCRIPTION:
Inclusion criteria：

1. Disease characteristics • Histologically confirmed rectal adenocarcinoma; Immunohistochemical confirmation as pMMR or/and pCR or/and NGS test as MSS;

   • Tumor location within 12cm from anal margin;
   * Locally advanced rectal cancer (stage II-III, i.e. cT3-4 and/or N+) as assessed by the UICC/AJCC TNM staging system (8th edition, 2017);

     * Preoperative staging method: pelvic MRI/ transrectal ultrasound combined with preoperative staging.
   * No signs of intestinal obstruction; Or intestinal obstruction has been relieved after proximal colostomy surgery;
   * Preoperative chest, abdominal and pelvic CT to exclude distant metastasis.
2. Patient characteristics

   • Age: 18 ~75 years old;
   * Activity status score: ECOG 0-1;
   * Life expectancy: more than 2 years;
   * Hematology: WBC>3500×106/L; PLT>100000×106/L; Hb>10g/dL;
   * Liver function: SGOT and SGPT are less than 1.5 times of normal value; Bilirubin less than 1.5mg/dL;
   * Kidney function: creatinine <1.8mg/dL;
   * Other: non-pregnant or breastfeeding women; No other malignant disease (other than non-melanoma or carcinoma in situ of the cervix) within 5 years or during the same period; Does not have a mental illness that prevents informed consent; There were no other serious diseases associated with shorter survival.
   * Patients or family members can understand the study protocol and are willing to participate in the study, and sign a written informed consent;
   * Good patient compliance, voluntary follow-up, treatment, laboratory tests, and other research steps as scheduled.
3. Prior treatment • No previous rectal cancer surgery;

   • No previous chemotherapy or radiation therapy;

   • No previous biotherapy;

   • Previous endocrine therapy: No restriction.

   Exclusion criteria：

   • CRC for microsatellite highly unstable (MSI-H) or mismatch repair protein expression deficiency (dMMR);

   • Chronic hepatitis B or C with a history or active HIV infection (high copy of viral DNA);

   • Autoimmune diseases;

   • Other active clinical serious infections (>NCI-CTC version 3.0);

   • Stage I patients;

   • Preoperative evidence of distant metastasis;

   • Dysfluid, organ function decompensation;

   • A history of pelvic or abdominal radiotherapy;
   * Multiple primary cancers;
   * Patients whose seizures require management (such as steroid or antiepileptic therapy);
   * A history of other malignancies within 5 years, except for cured cervical carcinoma insitu or skin basal cell carcinoma;
   * Chronic inflammatory bowel disease, intestinal obstruction; Substance abuse and medical, psychological or social conditions that may interfere with the patient's participation in the study or the evaluation of the findings;
   * A known or suspected allergy to the study drug or to any drug administered in connection with this trial;
   * Any unstable conditions or conditions that could compromise patient safety and compliance;

   Describe the medication or treatment in detail:

   1.1 Induction therapy stage (2 cycles of chemotherapy combined with immunotherapy)

1 Envafolimab: 200mg, subcutaneous injection, Q2W, 2 cycles (simultaneous administration on the first day of chemotherapy).

2mFOLFOX6: Q2W, 2 cycles: oxaliplatin 85mg/m2 intravenous infusion for 2h, day 1. Calcium folinate 400mg/m2 intravenous infusion for 2 hours, day 1. Fluorouracil was injected intravenously at 400mg/m2 on day 1, followed by 1200mg/ (m2·d) × 2d with continuous intravenous infusion (total 2400mg/m2, infusion for 46~48h). 1.2 Simultaneous chemoradiotherapy (long-term radiotherapy

Chemotherapy combined with immunotherapy for 3 cycles)

Radiation therapy: 50Gy/25f, 2Gy daily, 5 days a week for 5 weeks.

Body position fixation: prone position, full bladder, body fixator or vacuum bag fixation;

CT scan: Before the scan, intravenous contrast agent was injected to develop the intestine, fill the bladder, empty the intestine, and collect two sets of CT images of plain scan and enhanced phase (only plain scan images can be collected for those allergic to contrast agent).

Radiotherapy equipment: linear accelerator;

Target area and irradiation field: The target area includes the primary rectal area and lymphatic drainage area. The treatment plan is designed by IMRT radiotherapy. The target area coverage and normal tissue limit are determined by the radiotherapy doctor according to the specific conditions of the patient.

2 Capecitabine: 825mg/m2 orally (1650mg/m2/d) twice a day in the morning and evening, 5 days a week, synchronized with radiation therapy, for a total of 25 days.

3 Envafolimab: 200mg, subcutaneous injection, Q2W, 3 cycles (given on day 1, day 15, day 29 of radiotherapy).

1.3 Consolidation treatment stage (2 cycles of chemotherapy combined with immunotherapy)

1. Envafolimab: 200mg, subcutaneous injection, Q2W, 2 cycles, synchronous administration on the first day of chemotherapy.
2. mFOLFOX6: Q2W, 2 cycles: oxaliplatin 85mg/m2 intravenous infusion for 2h, day 1. Calcium folinate 400mg/m2 intravenous infusion for 2 hours, day 1. Fluorouracil was injected intravenously at 400mg/m2 on day 1, followed by 1200mg/ (m2·d) ×2d with continuous intravenous infusion (total 2400mg/m2, infusion for 46~48h).

ELIGIBILITY:
Inclusion Criteria:

* 1) Disease characteristics

  * Histologically confirmed rectal adenocarcinoma; Immunohistochemical confirmation as pMMR or/and pCR or/and NGS test as MSS;
  * Tumor location within 12cm from anal margin;
  * Locally advanced rectal cancer (stage II-III, i.e. cT3-4 and/or N+) as assessed by the UICC/AJCC TNM staging system (8th edition, 2017);

    * Preoperative staging method: pelvic MRI/ transrectal ultrasound combined with preoperative staging.
  * No signs of intestinal obstruction; Or intestinal obstruction has been relieved after proximal colostomy surgery;
  * Preoperative chest, abdominal and pelvic CT to exclude distant metastasis. 2) Patient characteristics
  * Age: 18 ~75 years old;
  * Activity status score: ECOG 0-1;
  * Life expectancy: more than 2 years;
  * Hematology: WBC>3500×106/L; PLT>100000×106/L; Hb>10g/dL;
  * Liver function: SGOT and SGPT are less than 1.5 times of normal value; Bilirubin less than 1.5mg/dL;
  * Kidney function: creatinine <1.8mg/dL;
  * Other: non-pregnant or breastfeeding women; No other malignant disease (other than non-melanoma or carcinoma in situ of the cervix) within 5 years or during the same period; Does not have a mental illness that prevents informed consent; There were no other serious diseases associated with shorter survival.
  * Patients or family members can understand the study protocol and are willing to participate in the study, and sign a written informed consent;
  * Good patient compliance, voluntary follow-up, treatment, laboratory tests, and other research steps as scheduled.

    3) Prior treatment
  * No previous rectal cancer surgery;
  * No previous chemotherapy or radiation therapy;
  * No previous biotherapy;
  * Previous endocrine therapy: No restriction.

Exclusion Criteria:

* CRC for microsatellite highly unstable (MSI-H) or mismatch repair protein expression deficiency (dMMR); Chronic hepatitis B or C with a history or active HIV infection (high copy of viral DNA);

  * Autoimmune diseases;
  * Other active clinical serious infections (>NCI-CTC version 3.0);
  * Stage I patients;
  * Preoperative evidence of distant metastasis;
  * Dysfluid, organ function decompensation;
  * A history of pelvic or abdominal radiotherapy;
  * Multiple primary cancers;
  * Patients whose seizures require management (such as steroid or antiepileptic therapy);
  * A history of other malignancies within 5 years, except for cured cervical carcinoma in situ or skin basal cell carcinoma;
  * Chronic inflammatory bowel disease, intestinal obstruction; Substance abuse and medical, psychological or social conditions that may interfere with the patient's participation in the study or the evaluation of the findings;
  * A known or suspected allergy to the study drug or to any drug administered in connection with this trial;
  * Any unstable conditions or conditions that may compromise patient safety and compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
pCR | 3 months
  Pathological complete response

SECONDARY OUTCOMES:
TRG | 3 months
  Pathological downphase rate

CONTACTS AND LOCATIONS:
Locations (1):
- Envafolimab, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT06239870/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT06239870/ICF_001.pdf